CLINICAL TRIAL: NCT00163852
Title: Salt Replacement for Metabolic Alkalosis in Acute Exacerbations of Cystic Fibrosis
Brief Title: Treatment of Metabolic Alkalosis in Acute Exacerbations of Cystic Fibrosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other); Monash University (Other); Cystic Fibrosis Federation Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Metabolic alkalosis; Hypercapnia; Salt replacement
MeSH Terms: conditions — Cystic Fibrosis; Hypercapnia | interventions — Salts

INTERVENTIONS:
Drug: Normal saline IV, salt tablets

SUMMARY:
Adult cystic fibrosis (CF) patients admitted with an acute infection complicated by acid-base disturbance and decreased ventilation will be studied.

They will receive salt replacement to correct the acid-base disturbance and possibly their ventilation.

Assessment of symptoms (questionnaire), acid-base and electrolyte status (blood and urine tests) ventilation (overnight oxygen and carbon dioxide monitoring non-invasively) and sleep-wake pattern (actigraphy) will be carried out.

Study hypothesis: Acute volume and electrolyte replacement corrects hypochloremic hypovolemic metabolic alkalosis and compensatory hypoventilation/ hypercapnia in acute exacerbations of cystic fibrosis.

DETAILED DESCRIPTION:
Background: Hypochloremic hypovolemic metabolic alkalosis contributes to hypercapnia in acute exacerbations of cystic fibrosis. Treatment of the metabolic alkalosis with volume and sodium chloride (NaCl) replacement could reduce hypoventilation and hypercapnia, thereby improving symptoms, sleep patterns and daytime activity level. This would avoid unnecessary treatment with non-invasive ventilation.

Hypothesis: Volume and NaCl replacement corrects hypochloremic hypovolemic metabolic alkalosis and compensatory hypoventilation/ hypercapnia in acute exacerbations of cystic fibrosis and results in symptomatic improvement.

Entry criteria:

* Adult cystic fibrosis patient
* Admission with acute exacerbation
* PaCO2 > 45 mmHg
* Primary metabolic alkalosis (acid-base diagram of Stinebaugh and Austin)
* Serum chloride (Cl) ≤ 98 mmol/L
* Serum albumin (alb) > 25 mmol/L

Intervention:

* Normal saline intravenously day(D)1,2,3. (Replace greater of Cl deficiency or acute weight loss, with 2/3 on D1 and remainder D2, D3)
* NaCl tablets 3 tds D4 to 10 (calculated to replace 7 mmol NaCl loss in 60 kg subject)

Random allocation to either:

1. Intervention + standard care (including standard dietary advice) D1-10
2. Standard care alone (including standard dietary advice) D1-10

Primary outcome measures: (D1, D4, D10)

* PaCO2 (performed at same time of day as admission ABG's)
* Acid-base status (Stinebaugh and Austin, ABG's)
* Serum chloride
* Overnight oximetry (% night SpO2<90%) and PtcCO2 (rise in CO2 overnight)

Secondary outcome measures: (D1, D4, D10)

* Serum albumin, sodium
* Body mass index (BMI)
* Spirometry (D1, D10)
* Headache scale
* Epworth sleepiness scale
* Wrist actigraphy (circadian rhythm and daytime activity level)(D1-10)
* Urinary chloride, potassium, sodium, pH, osmolality
* Baseline ABG's as stable outpatient (within 3 months, pre or post admission)

ELIGIBILITY:
Inclusion Criteria:

* Adult cystic fibrosis patient
* Admission with acute exacerbation (criteria- fall in FEV1 > 10% from best in last 12/12, change in sputum volume and colour, new pulmonary infiltrate)
* PaCO2 > 45 mmHg on admission
* Primary metabolic alkalosis (acid-base diagram of Stinebaugh and Austin)
* Serum chloride (Cl) ≤ 98 mmol/L
* Serum albumin (alb) ≤ 25 mmol/L

Exclusion Criteria:

Concurrent diuretic therapy Concurrent glucocorticoid therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2006-02

PRIMARY OUTCOMES:
Primary outcome measures: (Day1, D4, D10)
•PaCO2 (performed at same time of day as admission ABG's)
•Acid-base status (Stinebaugh and Austin, ABG's)
•Serum chloride
•Overnight oximetry (% night SpO2<90%) and PtcCO2 (rise in CO2 overnight)

SECONDARY OUTCOMES:
Secondary outcome measures: (Day1, D4, D10)
•Serum albumin, sodium
•Body mass index (BMI)
•Spirometry (D1, D10)
•Headache scale
•Epworth sleepiness scale
•Wrist actigraphy (circadian rhythm and daytime activity level)(D1-10)
•Urinary chloride, potassium, sodium, pH, osmolality
•Baseline ABG's as stable outpatient (within 3 months, pre or post admission)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Naughton, MBBS, MD, Principal Investigator — The Alfred
Locations (1):
- The Alfred, Melbourne, Victoria, Australia